CLINICAL TRIAL: NCT05371379
Title: A Multiple-dose, Randomized, Double Blind, Placebo-controlled, Dose-escalation Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of CM338 Injection in Healthy Subjects
Brief Title: Multiple Ascending Dose Study of CM338 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM338-100002
Record Dates: First submitted 2022-05-07; First posted 2022-05-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CM338 75 mg, subcutaneous injection (Experimental): Qquaque week
  Interventions: Biological: CM338 Injection
- CM338 150 mg, subcutaneous injection (Experimental): Qquaque week
  Interventions: Biological: CM338 Injection
- CM338 300 mg, subcutaneous injection (Experimental): Qquaque week
  Interventions: Biological: CM338 Injection
- CM338 300 mg, intravenous infusion (Experimental): Qquaque week
  Interventions: Biological: CM338 Injection
- Placebo (Placebo Comparator): placebo
  Interventions: Biological: CM338 Injection

INTERVENTIONS:
Biological: CM338 Injection — A humanized monoclonal antibody.

SUMMARY:
This study was a multi-center, randomized, double blind, placebo-controlled, single-dose, dose escalation Phase I study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of CM338 with multiple dosing in healthy subjects.

DETAILED DESCRIPTION:
The study included screening period, administration and safety follow-up period.

Forty-eight healthy volunteers will be enrolled and randomized into 4 groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, aged ≥18 and ≤65 years.
* Medical history, vital signs, physical examination, 12-lead ECG, X-ray, and abdominal color ultrasound results are normal, or abnormal without clinically significance.
* All clinical laboratory examination are normal, or abnormal without clinical significance.

Exclusion Criteria:

* Take any prescription medicine within 2 weeks before administration, or take any Chinese medicine or non-prescription medicine within 1 week.
* Live attenuated vaccine was administered within 30 days prior to administration or planned to vaccinate during the study period.
* Major surgery will be planned during the study period, or major surgery was performed within 4 weeks prior to dosing.
* Any blood loss greater than 400 mL by voluntary blood donation or in any other manner within 4 weeks prior to administration.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs). | Up to Week 12.
  Incidence of AEs, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.

CONTACTS AND LOCATIONS:
Locations (1):
- PKUCare Luzhong Hospital, Zibo, China